CLINICAL TRIAL: NCT05511792
Title: Transcatheter Aortic Valve Replacement For Patients With Bicuspid Aortic Stenosis (Type 0) Using Down Sizing Strategy Compared With Standard Sizing Strategy (HANGZHOU Solution): A Prospective, Multicenter, Randomized Controlled Trial
Brief Title: Down Sizing Strategy (HANGZHOU Solution) vs Standard Sizing Strategy TAVR in Bicuspid Aortic Stenosis (Type 0)
Acronym: TAILOR-TAVR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SAHZU 2022-0327
Record Dates: First submitted 2022-06-28; First posted 2022-08-23 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Aortic Stenosis With Bicuspid Valve

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants and Outcomes Assessors all remain unaware of the intervention assignments throughout the trial.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- TAVR with down sizing strategy (Experimental): Balloon sizing will be used during procedural. Pre-dilation with balloon size just below the annular size. 20mm for annular size of 20-23mm. 23mm for annular size 23-26mm.
  Waist sign with less than mild contrast regurgitation: Evolut PRO Valve one size smaller than manufacturer recommendation and Target implant depth 0-3mm.
  No waist sign and/or contrast regurgitation or unable to finish supra-annular sizing: Evolut PRO annular sizing (per manufacturer recommendation) with implant depth 0-3mm.
  Interventions: Procedure: TAVR for BAV Using Down Sizing with the Evolut Pro platform
- TAVR with standard sizing strategy (Active Comparator): Pre-dilation with balloon size just below the annular size. 20mm for annular size of 20-23mm. 23mm for annular size 23-26mm.
  The prosthesis size of Evolut PRO will be chosen based on manufacturer recommendation. The target implant depth will be 0-3mm.
  Interventions: Procedure: TAVR for BAV Using Traditional Sizing strategy with the Evolut Pro platform

INTERVENTIONS:
Procedure: TAVR for BAV Using Down Sizing with the Evolut Pro platform — Down sizing strategy in Type 0 bicuspid aortic stenosis patients undergoing transcatheter aortic valve replacement with self-expanding valves
  Other Names: Down Sizing Strategy
  Arms: TAVR with down sizing strategy
Procedure: TAVR for BAV Using Traditional Sizing strategy with the Evolut Pro platform — Traditional sizing strategy in Type 0 bicuspid aortic stenosis patients undergoing transcatheter aortic valve replacement with self-expanding valves
  Other Names: Standard Sizing Strategy
  Arms: TAVR with standard sizing strategy

SUMMARY:
To compare down sizing strategy versus annular sizing strategy technique (control group) in Type 0 bicuspid aortic stenosis (AS) patients undergoing transcatheter aortic valve replacement (TAVR) with self-expanding valves (SEVs): a randomized superiority trial

DETAILED DESCRIPTION:
Transcatheter aortic valve replacement (TAVR) has emerged as a favorable alternative for severe symptomatic aortic stenosis (AS) patients of all surgical risk profiles. Patients with bicuspid aortic valve (BAV) underwent TAVR had similar 30-day mortality as well as stroke and new pacemaker implantation rates compared to tricuspid aortic valve (TAV) subjects, but carried higher risk of moderate/severe perivalvular leakage (PVL), conversion to surgery and device failure. Clinical experience in China suggests BAV and heavy calcium burden are more common among TAVR candidates than US/EU cohorts.

Morphological characteristics at supra-annular structure (from annulus to the level of sinotubular junction) are quite complex in BAV, especially concomitant with heavily calcified leaflets. From our previous single center clinical practice, "waist sign" above the annulus during balloon aortic valvuloplasty in TAVR was often observed in patients with bicuspid AS, suggesting that supra-annular structures are the most constrained portion of BAV anatomy where the prosthesis anchors and seals. Therefore, we developed a balloon based supra-annular sizing strategy for self-expanding valves implantation in BAV and the device failure rate as well as pacemaker implantation rates were relatively low as shown in previous cohort study. Several other studies have also achieved successful outcomes associated with device "down sizing" (using a device smaller than that recommended by annular sizing).

The aim of this study is to compare "down sizing"strategy (experimental group) versus annular sizing strategy (control group) in BAV patients undergoing TAVR with self-expanding valves.

ELIGIBILITY:
Inclusion criteria:

1. Age ≥ 65 years;
2. Age <65 years and age ≥ 60 years with high surgical risk after combing STS Risk Estimate (≥ 8%), Katz activities of Daily Living, major Organ System Dysfunction and Procedure-Specific Impediment;
3. Severe, bicuspid aortic stenosis: Mean gradient ≥40 mmHg OR Maximal aortic valve velocity ≥4.0 m/sec OR Aortic valve area ≤1.0 cm2 (or aortic valve area index of ≤0.6 cm2/m2); if SVi <35mL/m2, low-dose dobutamine stress echocardiography is required;
4. NYHA classification ≥ II;
5. Type 0 (Sievers classification) by MDCT;
6. Perimeter-derived annulus diameter ranges from 20.0 mm to 26.0 mm;
7. Candidate for Transfemoral TAVR;
8. The study patient has been informed of the nature of the study, agrees to its provisions and has provided written informed consent as approved by the Institutional Review Board (IRB)/Ethics Committee (EC) of the respective clinical site.

Exclusion Criteria:

1. Any contra-indication for Self-expanding bioprosthetic aortic valve deployment Leukopenia (WBC < 3000 cell/mL), acute anemia (Hgb < 9 g/dL), Thrombocytopenia (Plt< 50,000 cell/mL).
2. Active sepsis, including active bacterial endocarditis with or without treatment;
3. Evidence of an acute myocardial infarction ≤ 1 month (30 days) before the intended treatment [(defined as: Q wave MI, or non-Q wave MI with total CK elevation of CK-MB ≥ twice normal in the presence of MB elevation and/or troponin level elevation (WHO definition)].
4. Stroke or transient ischemic attack (TIA) within 3 months (90 days) of the procedure.
5. Estimated life expectancy < 12 months (365 days) due to carcinomas, chronic liver disease, chronic renal disease or chronic end stage pulmonary disease.
6. Any Emergent surgery required before TAVR procedure.
7. A known hypersensitivity or contraindication to any of the following that cannot be adequately medicated:aspirin or heparin (HIT/HITTS) and bivalirudin; clopidogrel; Nitinol (titanium or nickel); contrast media
8. Gastrointestinal (GI) bleeding that would preclude anticoagulation.
9. Subject refuses a blood transfusion.
10. Severe dementia (resulting in either inability to provide informed consent for the study/procedure, prevents independent lifestyle outside of a chronic care facility, or will fundamentally complicate rehabilitation from the procedure or compliance with follow-up visits).
11. Other medical, social, or psychological conditions that in the opinion of the investigator precludes the subject from appropriate consent or adherence to the protocol required follow-up exams.
12. Currently participating in an investigational drug or another device study (excluding registries).
13. Hypertrophic cardiomyopathy (HCM with myocardium more than 1.5cm without an identifiable cause) with obstruction (HOCM).
14. Echocardiographic evidence of intracardiac mass, thrombus or vegetation.
15. Severe mitral stenosis amenable to surgical replacement or repair.
16. Aortic valve type cannot be determined (Sievers classification).
17. Significant aortic disease, including marked tortuosity (hyperacute bend), aortic arch atheroma [especially if thick (> 5 mm), protruding or ulcerated] or narrowing (especially with calcification and surface irregularities) of the abdominal or thoracic aorta, severe"unfolding" and horizontal aorta(Annular Angulation>70°).
18. Ascending aorta diameter > 50 mm.
19. Aortic or iliofemoral vessel characteristics that would preclude safe placement of the introducer sheath.
20. Patient is considered high risk for TAVR by CT corelab, including coronary obstruction, annular rupture and other severe TAVR-Related complications.
21. Previous pacemaker implantation.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 206 (Estimated)
Dates: Start 2022-06-27 (Actual); Primary Completion 2026-07-30 (Estimated); Study Completion 2030-06-30 (Estimated)

PRIMARY OUTCOMES:
Composite endpoint of Clinical Event Rate of Device Success (VARC-3), Free of pacemaker implantation, and Free of new onset complete left bundle branch block at 1 month | 1 month after index procedure
  Composite endpoint of Device Success (VARC-3), Free of pacemaker implantation, and Free of new onset complete left bundle branch block at 1 month

SECONDARY OUTCOMES:
New onset complete left bundle branch block | 1 month after index procedure
  New onset complete left bundle branch block with QRS ≥120ms at 1 month
Permanent pacemaker implantation | 1 month after index procedure
  Permanent pacemaker implantation within one month
Device success Rate | 1 month after index procedure
  Device success per VARC-3 definition
More than (≥) moderate regurgitation | 1 month after index procedure
  More than (≥) moderate regurgitation on echocardiography at 1month

CONTACTS AND LOCATIONS:
Overall Officials: Jian' an Wang, PhD, MD, Study Chair — 2nd Affiliated Hospital, School of Medicine, Zhejiang University, China
Locations (15):
- China (15):
  - Fujian Provincial Hospital, Affiliated to Fuzhou University, Fuzhou, Fujian
  - Xiamen Cardiovascular Hospital Xiamen University, Xiamen, Fujian
  - Lanzhou University First Hospital, Lanzhou, Gansu
  - Nanfang Hospital of Southern Medical University, Guangzhou, Guangdong
  - SUN YAT-SEN MEMORIAL HOSPITAL SUN YAT-SEN University, Guangzhou, Guangdong
  - Yulin First People's Hospital, Yulin, Guangxi
  - Zhengzhou Seventh People's Hospital, Zhengzhou, Henan
  - The Second XIANGYA Hospital Of Central South University, Changsha, Hunan
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - First Affiliated Hospital of Xi 'an Jiaotong University, Xi'an, Shaanxi
  - Affiliated Hospital of Qingdao University, Qingdao, Shandong
  - Qingdao Municipal Hospital, Qingdao, Shandong
  - Xinjiang Uygur Autonomous Region People's Hospital, Ürümqi, Xinjiang
  - The Second Affiliated Hospital Zhejiang University School of Medicine., Hangzhou, Zhejiang
  - Ning Bo First Hospital, Ningbo, Zhejiang

IPD SHARING:
Plan to Share IPD: No
undecided

REFERENCES:
- [Derived] Guo Y, Liu X, Li R, Ng S, Liu Q, Wang L, Hu P, Ren K, Jiang J, Fan J, He Y, Zhu Q, Lin X, Li H, Wang J. Comparison of downsizing strategy (HANGZHOU Solution) and standard annulus sizing strategy in type 0 bicuspid aortic stenosis patients undergoing transcatheter aortic valve replacement: Rationale and design of a randomized clinical trial. Am Heart J. 2024 Aug;274:65-74. doi: 10.1016/j.ahj.2024.04.011. Epub 2024 May 1. PMID 38701961